CLINICAL TRIAL: NCT01962480
Title: The Clinical Effects of Intracorporally Closure of the Hernia Defect in Laparoscopic Umbilical or Epigastric Hernia Repair
Brief Title: The Effect of Laparoscopically Closing the Hernia Defect in Laparoscopic Ventral Hernia Repair on Postoperative Pain
Acronym: CLOSE-GAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Mette Willaume Christoffersen, M.D, PhD, Hvidovre University Hospital
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLOSE-GAP-1
Record Dates: First submitted 2013-10-07; First posted 2013-10-14 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Ventral Hernias
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sutured closure of the hernia gap (Active Comparator): The hernia gap is sutured intracorporally
  Interventions: Procedure: The hernia gap is sutured intracorporally
- No closure of the hernia gap (No Intervention): Physiomesh is placed with at least 5 cm overlap of the gap and fixated with double crown technique

INTERVENTIONS:
Procedure: The hernia gap is sutured intracorporally — The hernia gab is closed with non-absorbable suture (Ethibond Excel 2-0, Ethicon, Johnson & Johnson©) performed by an intracorporally interrupted sutured technique using an Auto Suture© Endo-Slide knot-tying instrument. The stitches are placed with a distance of 0.5 - 1 cm from the fascial edges and with a distance of 0.5-1 cm. between the stitches, performed under a 6-8 mmHg intrabdominal pressure.
  Arms: sutured closure of the hernia gap

SUMMARY:
Introduction: Closure of the hernia gap in laparoscopic ventral hernia repair before mesh reinforcement has gained increasing acceptance among surgeons despite creating a tension-based repair. Beneficial effects of this technique have sporadically been reported but no evidence is available from randomized controlled trials.

The primary purpose is to compare early postoperative activity-related pain in patients undergoing ventral hernia repair with closure of the gap with patients undergoing standard laparoscopic ventral hernia repair (non-closure of the gap). Secondary outcomes are cosmesis and hernia-related quality of life (QoL) at 30-days and clinical or radiological recurrence and chronic pain after 2 years.

Material and Methods: A randomized, controlled, double-blinded study is planned. Based on power calculation we will include 40 patients in each arm. Patients undergoing elective laparoscopic umbilical, epigastric, or umbilical trocar-site hernia repair at Hvidovre Hospital, Herlev Hospital, or Køge Hospital, who meet the inclusion criteria, are invited to participate.

Conclusion: The technique with closure of the gap may induce more postoperative pain, but may be superior with regard to other important surgical outcomes. No studies have previously investigated closure of the gap in the setting of a randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria
* Elective, primary or recurrent laparoscopic umbilical or epigastric hernia repair, umbilical trocar-site hernia and epigastric hernia repair where laparoscopic hernia repair is no contraindication (i.e. previous laparotomy with anticipated severe and dense adhesions
* Hernia defect between 2-6 cm measured preoperatively by the surgeon at the out-patient clinic
* Maximum 1 defect
* Patients 18-80 years Patients with technical failure (where it is not possible to suture the defect) or patients who are reoperated due to complications remain included and will stay in their primary assigned randomization group in order to perform an intention to treat (ITT) analysis.

Exclusion Criteria:

* Open hernia repair
* Poor compliance (language problems, dementia and alcohol or drug abuse etc.)
* Fascia defect >6 cm (largest diameter, evaluated preoperatively and intra-operatively, thus patients are excluded if the defect is found larger intra-operatively)
* Emergency repair
* Chronic pain syndrome (chronic back pain, chronic headache, severe dysmenorrhea, fibromyalgia, whiplash or other conditions requiring daily opioid medication)
* Daily consumption of opioids (for the last 3 weeks up till the operation)
* Decompensated liver cirrhosis (Child-Pugh B-C)
* If the hernia repair is secondarily to another surgical procedure
* If a patient withdraws his/her inclusion consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-11; Primary Completion 2016-08 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Pain at mobilisation from lying to sitting position measured with Visual Analogue Scale | 24 hrs postoperatively

SECONDARY OUTCOMES:
Cosmetic result measured with verbal rating scale and numeric rating scales | measured 30 days postoperatively

OTHER OUTCOMES:
Hernia-specific quality of life | measured 30 days postoperatively
  Measured with Carolina Comfort Scale (CCS)
complications, readmittance, and general practitioner visits | 30-days postoperatively
  Measured with patient interview, and/or patient files
clinical recurrence | 2 years
  clinical or radiological recurrence
chronic pain | within 2 years
  moderate or severe chronic pain after 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mette Christoffersen, M.D., Principal Investigator — Individual Purchaser
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sauerland S, Walgenbach M, Habermalz B, Seiler CM, Miserez M. Laparoscopic versus open surgical techniques for ventral or incisional hernia repair. Cochrane Database Syst Rev. 2011 Mar 16;(3):CD007781. doi: 10.1002/14651858.CD007781.pub2. PMID 21412910
- [Derived] Christoffersen MW, Westen M, Rosenberg J, Helgstrand F, Bisgaard T. Closure of the fascial defect during laparoscopic umbilical hernia repair: a randomized clinical trial. Br J Surg. 2020 Feb;107(3):200-208. doi: 10.1002/bjs.11490. PMID 31971616
- [Derived] Christoffersen MW, Westen M, Assadzadeh S, Deigaard SL, Rosenberg J, Bisgaard T. The clinical effects of closure of the hernia gap after laparoscopic ventral hernia repair: protocol for a randomised controlled trial. Dan Med J. 2014 Jun;61(6):A4865. PMID 24947633